CLINICAL TRIAL: NCT05070663
Title: National, Multicentre, Non-interventional, Prospective and Retrospective Study in Adolescent Patients With Severe Uncontrolled Asthma Starting Treatment With Dupilumab (Dupixent®)
Brief Title: A Study in Male and Female Adolescent Participants With Severe Uncontrolled Asthma Starting Treatment With Dupilumab Injection (Dupixent®)
Acronym: PEDIASTHMA
Status: Completed | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS17083; U1111-1256-9593 (Registry Identifier: ICTRP)
Record Dates: First submitted 2021-09-27; First posted 2021-10-07 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 52 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants with severe asthma: Adolescents, for whom initiation of dupilumab (Dupixent®) for the severe uncontrolled asthma indication was decided by the investigator before the inclusion in the study.

SUMMARY:
Primary objective:

- Describe the characteristics of enrolled severe asthma patients

Secondary objectives:

* Assess the control of asthma under dupilumab (Dupixent®) treatment until 1 year
* Assess the clinical objectives of the asthma care
* Assess comorbidities associated with Type 2 inflammation
* Assess safety during the year of treatment

DETAILED DESCRIPTION:
52 weeks

ELIGIBILITY:
Inclusion Criteria:

* Adolescents, for whom initiation of dupilumab (Dupixent®) for the severe uncontrolled asthma indication was decided by the investigator before the inclusion in the study
* Adolescents ≥ 12 and < 18 years of age at the time of the initiation of Dupixent® treatment

Exclusion Criteria:

- Adult participants ≥ 18 years of age

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescents, for whom initiation of dupilumab (Dupixent®) for the severe uncontrolled asthma indication was decided by the investigator before the inclusion in the study.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Medical history (including history of asthma) | At the start of treatment with Dupixent® (day 1)
  Relevant medical history other than asthma according to the investigator (including documented comorbidities associated with type 2 inflammation). Asthma history includes patient age at the time of diagnosis and family history.
Previous treatments for asthma | At the start of treatment with Dupixent® (day 1)
  Background asthma treatments (doses and international nonproprietary name (INN) of inhaled corticosteroids (ICS), long-acting beta-2 agonist (LABA) and oral corticosteroids (OCS), etc) including cumulative yearly dose of OCS. Use of oral corticosteroids due to exacerbation of asthma (dose, INN). Use of emergency treatments (short-acting beta-2 agonist (SABA)) (number of times per week).
Demographic characteristics | At the start of treatment with Dupixent® (day 1)
  Age and gender.
Disease characteristics | At the start of treatment with Dupixent® (day 1)
  Disease characteristics at the inclusion including severity (Global Initiative for Asthma (GINA) step), number of severe exacerbations during the past year, number of days in intensive care unit (ICU) for severe exacerbation since the diagnosis, forced expiratory volume per second (FEV1), Asthma Control Test (ACT) score.
Concomitant medication | At the start of treatment with Dupixent® (day 1)
  Relevant concomitant medication other than medication for asthma according to the investigator.

SECONDARY OUTCOMES:
Change from baseline to week 52 in asthma control test (ACT) score at each subsequent visit over the year of treatment | From baseline (day 1) to week 52
  ACT score range: 5-25; higher score indicates better asthma control.
Change from baseline to week 52 in number of annualized exacerbations and description of exacerbation setting | From baseline (day 1) to week 52
  An exacerbation is defined as deterioration of asthma requiring use of systemic corticosteroids for ≥3 days; or increase in oral corticosteroids (OCS) dose at ≥2 times the current dose for ≥3 days; or hospitalization or emergency room visit because of asthma, requiring systemic corticosteroids.
Change from baseline to week 52 in Paediatric Asthma Quality of Life Questionnaire (PAQLQ) score | From baseline (day 1) to week 52
  Questionnaire including 23 questions in 3 domains (symptoms, activity limitation, emotional function) and a 7-point scale (7 = not bothered at all; 1 = extremely bothered).
Change from baseline to week 52 in corticosteroid dose | From baseline (day 1) to week 52
  Change in corticosteroid dose.
Change from baseline to week 52 in pre- bronchodilator forced expiratory volume per second (FEV1) | From baseline (day 1) to week 52
  FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline to week 52 in number of food allergic reactions | From baseline (day 1) to week 52
  Following food allergic reactions will be recorded: allergic symptoms and anaphylaxis in real life or during an oral food challenge.
Change from baseline to week 52 in in visual analogue scale (VAS) score for allergic rhinitis | From baseline (day 1) to week 52
  VAS score range: 0 ('no symptoms') to 100 ('severe symptoms').
Change from baseline to week 52 in in Score for atopic dermatitis (SCORAD) score for atopic dermatitis | From baseline (day 1) to week 52
  SCORAD is a clinical tool for assessing the severity (i.e., extent, intensity) of atopic dermatitis as objectively as possible with scores ranging from 0-100. The higher the score indicates more severe atopic dermatitis.
Change from baseline to week 52 in sinonasal symptoms of nasal polyposis of food allergies | From baseline (day 1) to week 52
  Following sinonasal symptoms will be recorded: nasal congestion, loss in smell, posterior nasal discharge, anterior nasal discharge.
Responder rates at week 52 for ACT (according to the minimal important difference (MID)) | At week 52
  A participant is defined as responder if he/she has a change from baseline of 3 points or more at week 52 on the ACT score. ACT score range: 5-25; higher score indicates better asthma control.
Responder rates at week 52 for PAQLQ (according to the MID)) | At week 52
  A participant is defined as responder if he/she has a change from baseline of 0.5 points or more at week 52 on the PAQLQ score. The PAQLQ(S) overall score is calculated by adding points of individual responses to all questions, with the higher scores indicating less impairment that is, a better quality of life. Questionnaire including 23 questions in 3 domains (symptoms, activity limitation, emotional function) and a 7-point scale (7 = not bothered at all; 1 = extremely bothered).
Reasons for Dupixent® discontinuation | Day 1 to week 52
  All reasons for treatment discontinuation.
Collection of adverse events | Day 1 to week 52
  Number of adverse events.
Collection of serious adverse events | Day 1 to week 52
  Number of serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational site France, France, France

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org